CLINICAL TRIAL: NCT04181294
Title: Time Limited Trials to Reduce Non-Beneficial Intensive Care Unit Treatments Among Critically-ill Patients With Advanced Medical Illnesses
Brief Title: Time Limited Trials to Reduce Non-Beneficial Intensive Care Unit Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Los Angeles Department of Health Services (Unknown); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Dong Chang, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 0311710100
Record Dates: First submitted 2019-10-31; First posted 2019-11-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2019-10

CONDITIONS: Critical Illness; Communication
Keywords: Palliative Care; Medical Futility; Intensive Care
MeSH Terms: conditions — Critical Illness; Communication

STUDY DESIGN:
Intervention Model Description: Pre- and post study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (Experimental): Baseline data on patient characteristics and outcomes will be collected for 4 months prior to intervention.
  Interventions: Behavioral: Usual practice
- Post-intervention (Experimental): The quality improvement intervention will be conducted sequentially at all 3 medical centers (LAC-USC, Olive View, and Harbor-UCLA Medical Centers). Data on patient characteristics and outcomes will be collected for 4 months after the intervention
  Interventions: Behavioral: Family meetings using time limited trials as default ICU communication and care planning approach

INTERVENTIONS:
Behavioral: Family meetings using time limited trials as default ICU communication and care planning approach — Providers will be trained using didactics, focus groups, and simulations using actors as family members. A TLT protocol and checklist will be used to facilitate family meetings. A coordinator will schedule family meetings. Routine feedback sessions will be held with the local champions.
  Arms: Post-intervention
Behavioral: Usual practice — Baseline practice of ICU communication and care planning
  Arms: Pre-intervention

SUMMARY:
Overutilization of intensive care unit (ICU) treatments among patients with advanced medical illnesses and poor prognosis places them at risk for prolonged suffering with minimal anticipated benefit. Improving communication and shared decision-making between providers and patients/family members represents an opportunity to reduce potentially non-beneficial treatments. Time limited trials (TLTs) are agreements between clinicians and patients/surrogate decision-makers to use medical therapies over a defined period of time to observe if patients improve or deteriorate according to agreed-upon clinical outcomes. The objective of this project is to examine whether a quality improvement intervention that uses protocoled time limited trials as the default ICU communication/care planning strategy for patients with advanced medical illnesses will decrease the duration and intensity of non-beneficial ICU treatments without changing hospital mortality.

DETAILED DESCRIPTION:
Invasive intensive care unit (ICU) treatments for patients with advanced medical illnesses and poor prognoses may prolong suffering with minimal benefit. Unfortunately, the quality of care planning and communication between clinicians and critically-ill patients/families in these situations are highly variable, frequently leading to over-utilization of invasive ICU treatments. Time limited trials (TLTs) are agreements between the clinicians and patients/decision-makers to use certain medical therapies over defined periods of time and evaluate whether patients improve or worsen according to pre-determined clinical parameters. For patients with advanced medical illnesses receiving aggressive ICU treatments, TLTs can promote effective dialogue, develop consensus in decision-making, and set rational boundaries to treatments based on patients' goals of care. The objective of our study is to examine whether a multi-component quality improvement strategy that uses protocoled time limited trials as the default ICU care planning approach for critically-ill patients with advanced medical illnesses will decrease duration and intensity of non-beneficial ICU care without changing hospital mortality.

This study will be conducted in medical ICUs of 3 public teaching hospitals in Los Angeles County. We will train clinicians to use protocol-enhanced TLTs as the default communication and care planning approach in patients with advanced medical illnesses who receive invasive ICU treatments. Eligible patients will be those considered by treating ICU physicians to be at high risk for non-beneficial treatments according to guidelines from the Society of Critical Care Medicine. ICU physicians will be trained to use the TLT protocol through a curriculum of didactic lectures, case discussions, and simulations utilizing actors as family members in role-playing scenarios. Family meetings will be schedule by trained care managers. The improvement strategy will be implemented sequentially in the 3 participating hospitals, and outcomes will be evaluated using a before-after study design.

Key process outcomes will include frequency, timing, and content of family meetings. The primary clinical outcome will be ICU length of stay. Secondary outcomes will include hospital length of stay, days receiving life-sustaining treatments (mechanical ventilation, vasopressors, and renal replacement therapy), number of attempts at cardiopulmonary resuscitation, frequency of invasive ICU procedures, and disposition from hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the medical ICU who are determined on admission by the treating ICU physicians to be at high risk for potentially non-beneficial treatments based on ICU Admission and Triage Guidelines from the Society of Critical Care Medicine

Exclusion Criteria:

* Patients who cannot communicate for themselves and do not have surrogate decision-makers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
ICU Length of Stay | 4 months
  ICU LOS will be collected using the electronic medical record

SECONDARY OUTCOMES:
Hospital Length of Stay | 4 months
  Hospital LOS will be collected using the electronic medical record
Days receiving life-sustaining ICU treatments | 4 months
  Total number of days receiving mechanical ventilation, vasopressor medications, and renal replacement therapy will be collected from the electronic health record
Use of invasive ICU procedures | 4 months
  Total number of central venous or arterial catheterizations, thoracenteses, paracenteses, lumbar punctures, endoscopies, and attempts at cardiopulmonary resuscitation will be collected using the electronic health record

OTHER OUTCOMES:
Key process measure: Family meetings | 4 months
  A convenience sample of family meetings will be examined to determine the proportion of meetings in which key decision-making components (discussion of medical issues, prognosis, risk/benefit of ICU treatments, patients' values and preferences, clinical markers of improvement, recommendations for next steps) were discussed

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Los Angeles County-University of Southern California Medical Center, Los Angeles, California
  - Olive View Medical Center, Sylmar, California
  - Harbor UCLA Medical Center, Torrance, California

REFERENCES:
- [Derived] Chang DW, Neville TH, Parrish J, Ewing L, Rico C, Jara L, Sim D, Tseng CH, van Zyl C, Storms AD, Kamangar N, Liebler JM, Lee MM, Yee HF Jr. Evaluation of Time-Limited Trials Among Critically Ill Patients With Advanced Medical Illnesses and Reduction of Nonbeneficial ICU Treatments. JAMA Intern Med. 2021 Jun 1;181(6):786-794. doi: 10.1001/jamainternmed.2021.1000. PMID 33843946